CLINICAL TRIAL: NCT02981979
Title: Comparison of the Efficacy and Safety of Leflunomide Versus Placebo Combined With Basic Prednisone Therapy in Patients With Active Takayasu Arteritis: a Randomized Double-blind Controlled Clinical Trial
Brief Title: Takayasu Arteritis Clinical Trial in China
Acronym: TACTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiang lindi (Other)
Responsible Party: Sponsor-Investigator, Jiang lindi, Chief of Department of Rheumatology, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016ZSLC-06
Record Dates: First submitted 2016-11-22; First posted 2016-12-05 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Takayasu Arteritis
Keywords: Takayasu Arteritis; Leflunomide
MeSH Terms: conditions — Takayasu Arteritis | interventions — Leflunomide; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants were assigned randomly (1:1) to treatment with LEF or placebo according to a computer-generated blocked randomization list. The randomization list, which assigns a unique randomization number to each treatment, was generated and kept sealed by a randomization administrator (independent of the trial conduct and data analysis). Randomization was masked to patients, investigators, clinical outcome monitors, project managers and statisticians. The packaging of the LEF and placebo was identical with labelled randomization number. For emergency use, investigators were given a sealed opaque envelope for each randomization number. If an envelope was opened, the time, date and reason for opening had to be recorded on the envelope and signed by the investigator. At the end of the trial, all envelopes were returned to the principal investigator unopened to confirm that masking had been maintained throughout the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leflunomide group (Active Comparator): For the first 24 weeks, patients in the LEF group were treated with prednisone (0.6mg/kg/d, p.o.) and LEF (20mg/d, p.o.). The initial dose of prednisone was maintained for 4 weeks and then tapered by 5.0 mg every 2 weeks. The tapering of prednisone dose was determined by the investigators based on their assessment of disease activity. Two investigators formulated a tapering plan for the same time. If there were differences between the 2 investigators' perspectives, a third experienced senior rheumatologist (Lindi Jiang) made the final decision. Once the prednisone dose was reduced to 10 mg/d, this dose was maintained to the end of week 52.
  By week 24, if clinical remission had been achieved, the patients proceeded to maintenance therapy with LEF (20 mg/day) from week 25. If the patient did not meet the criteria for clinical remission, unblinding was carried out: patients in the LEF group discontinued the study.
  Interventions: Drug: Leflunomide(LEF); Drug: Prednisone Acetate Tablets
- Control Group (Placebo Comparator): For the first 24 weeks, patients in the placebo group received prednisone (0.6mg/kg/d, p.o.) and LEF simulator (2 tablets/d, p.o.). Patients were instructed to take tablets regularly. The initial dose of prednisone was maintained for 4 weeks and then tapered by 5.0 mg every 2 weeks. The tapering of prednisone dose was determined by the investigators based on their assessment of disease activity. Two investigators formulated a tapering plan for the same time. If there were differences between the 2 investigators' perspectives, a third experienced senior rheumatologist (Lindi Jiang) made the final decision. Once the prednisone dose was reduced to 10 mg/d, this dose was maintained to the end of week 52.
  By week 24, if clinical remission had been achieved, the patients proceeded to maintenance therapy with LEF (20 mg/day) from week 25. If the patient did not meet the criteria for clinical remission, unblinding was carried out: patients in the placebo group switched to LEF (20 mg/day) .
  Interventions: Drug: Leflunomide(LEF); Drug: Prednisone Acetate Tablets; Drug: Placebos

INTERVENTIONS:
Drug: Leflunomide(LEF) — Leflunomide:
  For LEF arm, 20mg per day, p.o. through the whole study. For placebo group, 20mg per day, p.o. from week 25 to week 52.
Drug: Prednisone Acetate Tablets — Prednisone (5mg/tab): basic therapy, start with 0.6mg/kg/d and maintained for 4 weeks, then reducing 5mg every 2 weeks until 10mg per day.
Drug: Placebos — 2 tabs/d used in placebo arm for the first 24 weeks.
  Arms: Control Group

SUMMARY:
To investigate the efficacy and safety of Leflunomide (LEF) versus placebo combined with prednisone for active Takayasu arteritis (TAK) in Chinese population.

DETAILED DESCRIPTION:
Takayasu arteritis (TAK) is a rare form of large-vessel vasculitis, characterized by immune -induced vascular inflammation, resulting in the stenosis and occlusion of blood vessels [1]. TAK is observed predominantly in Asian females under 40 years of age [2, 3]. The stenosis or occlusion of blood vessels can cause severe ischemic events (e.g., acute myocardial infarction, stroke, death) involving multiple organs. Patients with TAK experience impaired quality of life [4] and face a significantly higher risk of death compared with that in the sex- and age-matched general population, with a standardized mortality ranging from 2.7 to 17.3 [5, 6, 7]. Thus, timely and efficacious treatment is important to improve the prognosis in such a young population.

Glucocorticoids (GCs) are the first-line therapy for active TAK [8, 9]. High-dose GCs are initially efficacious. However, disease recurrence can occur in approximately 60% patients during the GCs tapering [10, 11]. Prolonged use of GCs is associated with significant toxicity, including glucose-metabolism disorders, cardiovascular adverse events (AEs), and osteoporosis [12, 13]. Therefore, immunosuppressive therapy is required to minimize the dose and duration of GC exposure [8, 9]. Conventional immunosuppressants have been recommended as GC-tapering agents for active TAK, whereas biological agents are recommended in refractory cases [8, 9]. Most previous studies focused on TAK treatment have been observational, only five randomized clinical trials (RCTs) are found, among which, just one study reported the effect of conventional immunosuppressants mycophenolate [14, 15, 16, 17, 18]. Thus, high-quality evidence to support therapeutic options of conventional immunosuppressants is very limited.

Leflunomide (LEF) is a conventional immunosuppressant [19], which has shown satisfied GC-tapering effects in the treatment of giant cell arteritis, another large vessel vasculitis, in several observational studies [20, 21, 22]. In 2012, the first open-label study of 14 TAK patients demonstrated that 70% of patients could achieve at least partial clinical remission, and the GC dose could be reduced by 50% during LEF treatment [23]. Since then, several observational cohort or case-control studies have reported the efficacy of LEF for active TAK [24, 25, 26, 27, 28, 29]. A most recent study reported a comparable complete response rate of LEF (78%) versus adalimumab (88%) at 15-month follow-up [30]. Thus, LEF would be a promising alternative treatment for TAK, but evidence from RCTs is lacking.

We conducted this multicenter, randomized, double-blind, placebo-controlled trial to investigate the efficacy and safety of LEF versus placebo combined with prednisone for active TAK, namely "Takayasu arteritis clinical trial in China" (TACTIC; ClinicalTrials.gov identifier: NCT02981979).

ELIGIBILITY:
Inclusion criteria i. Male or females aged 18-65 years diagnosed with TAK according to the classification criteria set by the American College of Rheumatology (ACR) in 1990; ii. With active disease within the last 3 months, meeting at least two of the following conditions:

1. new vascular ischemic manifestations/physical signs or systemic symptoms;
2. evaluated erythrocyte sedimentation rate (ESR) or high-sensitivity C reactive protein (hs-CRP) ≥6 mg/L or C reactive protein (CRP) ≥10 mg/L without other confounding factors (e.g., infection);
3. active vascular inflammation as indicated by contrast-enhanced computed tomography angiography (CTA), magnetic resonance angiography (MRA), color Doppler ultrasonography or positron emission tomography/CT (PET/CT); iii. Individuals should not receive LEF within 3 months before screening; iv. For individuals who received cyclophosphamide before screening, cyclophosphamide should be discontinued for ≥8 weeks; for patients who received a biological agent before screening, biological agents (e.g., tocilizumab, rituximab, and inhibitors of tumor necrosis factor) should be discontinued for ≥12 weeks; v. For patients who were taking prednisone (or its equivalent) before screening, the dose should be ≤0.6 mg/kg/day and the dose should be stable for ≥4 weeks; vi. Pregnancy should not be planned and a pregnancy test should be negative.

Exclusion criteria i. Individuals who had only vascular dilatation or aneurysm formation; ii. Individuals who had received revascularization surgery within the previous 3 months; iii. Individuals with severe organ dysfunction meeting at least one of the following:

1. heart dysfunction: New York Heart Association grade IV;
2. renal dysfunction: estimated glomerular filtration rate ≤60 mL/min;
3. liver dysfunction: Child-Pugh grade ≥2;
4. neurologic severe ischemic event: amaurosis on 3 consecutive days, acute cerebral infarction, or cerebral hemorrhage;
5. uncontrolled blood pressure >160/100 mmHg; iv. Individuals had at least one following abnormal laboratory test results:

(1) alanine aminotransferase or aspartate transaminase ≥1.5-fold of the upper limit of normal in serum; (2) white blood cell count ≤4×109/L; (3) platelet count ≤100×109/L; (4) hemoglobin ≤85 g/L; v. Individuals had other types of autoimmune disease or uncontrolled asthma who need prednisone ≥10 mg/day, a history of malignant tumor or any serious acute/chronic infection, including positivity for hepatitis B surface antigen, hepatitis C antibody, or clinical/radiological/laboratory evidence of active tuberculosis; vi. Individuals who were allergic to any of the investigational drugs; vii. Individuals had at least one of the following unacceptable treatments or medications:

1. previous treatment with LEF for ≥3 months but not efficacious;
2. planning to receive an attenuated vaccine during the study period;
3. planning to undergo (or have undergone) organ transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Achievement of clinical remission at week 24 | From the date of randomization until the end of induced remission therapy, assessed up to 24 weeks
  Clinical remission is defined as follows:
  (i) have no systemic symptoms (e.g., fever, fatigue, weight loss); (ii) have no new onset of ischemic symptoms and signs; (iii) have a normal level of erythrocyte sedimentation rate (ESR). If not achieved, the investigator excluded other influencing factors (especially infection), re-measure the ESR after 1 week, and use the re-examined value in the analyses.
  Subject achieving clinical remission should meet all these criteria above.
  The clinical remission rate and its difference between LEF and placebo group with 95% confidence interval (CI) at week 24 was estimated by Newcombe-Wilson procedure. If the lower limit of the 95%CI of the difference >10%, it is considered that the efficacy of LEF is significantly superior to placebo.

SECONDARY OUTCOMES:
Time to clinical remission | From the date of randomization until the date of first documented clinical remission, assessed up to 24 weeks
The mean prednisone dose at week 24 | At the end of induced remission therapy, assessed up to 24 weeks
Achievement of clinical remission at week 52 in those who switched from placebo to LEF from week 25 | From the time of switch from placebo to LEF treatment (week 25), assessed up to week 52
Disease recurrence through week 25 to week 52 | From the beginning of week 25 to the end of follow up, assessed up to week 52
  Disease recurrence is defined as NIH score ≥2 or not meeting ≥2 criteria for clinical remission.
  NIH score:
  1) presence of systemic symptoms as fever, fatigue and weight loss (1');
  2）presence of ischemic symptoms or signs (1');
  3) abnormal serum ESR levels (1');
  4) progression or new site of vascular lesions on MRA or CTA compared to baseline(1').
Time to recurrence | from the beginning of achieving clinical remission to the date of the first documented disease recurrence, assessed up to 52 weeks
Imaging changes at the end of week 24 and week 52 compared to the baseline | From the date of randomization until the end of week 24 and week 52
Safety-adverse events | From the date of randomization until the end of this trial, assessed up to 52 weeks
  For safety analysis, the incidence and severity of AEs, adverse drug reactions and laboratory values in the LEF and placebo group would be estimated and compared using the χ2 test or Fisher's exact test. The association of an abnormal laboratory index and adverse event with the investigational drug would be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, Doctor, Study Director — Fudan University
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Urumqi, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Wu B, Zhang W, Ma L, Kong X, Chen H, Jiang L. Comparison of the efficacy and safety of leflunomide versus placebo combined with basic prednisone therapy in patients with active disease phase of Takayasu arteritis: study protocol for a randomized, double-blinded controlled trial (Takayasu arteritis clinical trial in China: TACTIC). Ther Adv Chronic Dis. 2023 Mar 4;14:20406223231158567. doi: 10.1177/20406223231158567. eCollection 2023. PMID 36895331